CLINICAL TRIAL: NCT02096835
Title: Transcutaneous Electrical Acupoint P6 Stimulation vs. Tropisetron Both in Combination With Dexamethasone to Prevent Postoperation Nausea and Vomiting in Women
Brief Title: Transcutaneous Electrical Acupoint Stimulation of P6 to Prevent Postoperation Nausea and Vomiting
Acronym: TEASP6PPONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Yu Yang, MD, MD., Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TEAS-PONV
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative nausea and vomiting; Transcutaneous electrical acupoint stimulation; Gynecological laparoscopic surgery; Tropisetron; Dexamethasone
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Tropisetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acustimulation (Experimental): Transcutaneous electrical acupoint stimulation (TEAS) starts 30 min before surgery and lasts until patient leaves the postanesthetic care unit.Dexamethasone 10mg i.v. after induction.
  Interventions: Device: Transcutaneous electrical acupoint stimulation; Drug: Dexamethasone
- Tropisetron (Active Comparator): Tropisetron 5mg iv. at the start of skin closure.Sham transcutaneous electrical acupoint stimulation.Dexamethasone 10mg i.v.after induction.
  Interventions: Device: Sham transcutaneous electrical acupoint stimulation; Drug: Tropisetron; Drug: Dexamethasone
- Control (Sham Comparator): Sham transcutaneous electrical acupoint stimulation. Dexamethasone 10mg i.v.after induction.
  Interventions: Device: Sham transcutaneous electrical acupoint stimulation; Drug: Dexamethasone

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — A surface electrode will be applied to the P6 acupoint on the dominant upper extremity, located approximately 3cm proximal to the distal wrist crease between the tendons of the flexor carpi radialis and the palmaris longus, and a negative surface electrode placed on the opposing dorsum aspect of the forearm.
  Other Names: TEAS; Electrical neuromuscular stimulation device,JNR-2
  Arms: Acustimulation
Device: Sham transcutaneous electrical acupoint stimulation — The same TEAS protocol will be applied unless silicone covers will be attached to both electrodes. The device will also be turned on during the procedure.
  Arms: Control; Tropisetron
Drug: Tropisetron — will be given at the start of skin closure
  Other Names: Tropisetron Hydrocloride Injection; Batch number:131001
  Arms: Tropisetron
Drug: Dexamethasone — will be given after induction

SUMMARY:
The purpose of this study is to access the effect of TEAS of P6 in the prevention of PONV in women scheduled for gynecologic laparoscopic surgery with general anesthesia.

DETAILED DESCRIPTION:
150 female patients, aged between 18 to 60 y, who are scheduled for elective gynecological laparoscopic surgery requiring general anesthesia, will be randomly allocated by a computer generated randomization table to acustimulation group (Group Acu), tropisetron group (Group Trp),or dexamethasone group (Group Dxm).

In Group Acu, a surface electrode will be applied in the induction room to the P6 acupoint 30 min before induction.An operator will set electric stimulating current at 1mA with frequency at 2 Hz, and gradually increased the current intensity to a little below discomfort threshold.The stimulation will be maintained until the patient is discharged from the post-anesthesia care unit (PACU). In Group Trp and Group Dxm, the same protocol will be applied unless silicone covers attached to both electrodes.

A standardized anesthetic protocol will be followed. After induction, dexamethasone 10mg i.v. will be given in all groups. All patients will receive intravenous lactated Ringer's solution based on calculated preoperative deficits, surgical procedure, and estimated intraoperative blood loss. Parecoxib 40mg i.v. during surgery and incision infiltration of 0.5% ropivacaine at the end of surgery will be used for post-operative analgesia. After surgery, analgetic therapy will continue with morphine upon patient's request.After extubation, patients will be transported to PACU and observed for no less than 30 min. Metoclopramide 10mg i.v. will be administered as a rescue therapy to any patient who experiences an episode of moderate or severe nausea, an episode of vomiting, and requests rescue medication.

At the start of skin closure, a prefilled syringe which contains 5 ml of a solution will be administered intravenously to the patient. It will contain either saline (Group Acu and Group Dxm) or tropisetron 5mg (Group Trp).The syringe with the drug will be prepared by a study coordinator according to group allocation.

The patients, the anesthesiologists, and the nursing staff shall be unaware of the group assignments.

An anesthesiologist and an anesthetic nurse, who are trained for the study and blinded to the randomization, will collect the data.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II
* aged between 18 to 60yr
* scheduled for elective gynecological laparoscopic surgery requiring general anesthesia

Exclusion Criteria:

* pregnancy or breastfeeding
* mental retardation
* psychiatric or neurological disease
* use of antiemetics, emetogenic drugs, opioids or glucocorticosteroids within 3 days prior to surgery
* known allergy to tropisetron or dexamethasone
* nausea and/or vomiting within 24 hr prior to surgery
* implantation of a cardiac pacemaker, cardioverter, or defibrillator
* any skin problem at the acupoint stimulation area

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, PhD, Study Chair — Department of Anesthesiology, North Institute of Huashan Hospital,Fudan University
Locations (1):
- Department of Anesthesiology, North Institute of Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yang XY, Xiao J, Chen YH, Wang ZT, Wang HL, He DH, Zhang J. Dexamethasone alone vs in combination with transcutaneous electrical acupoint stimulation or tropisetron for prevention of postoperative nausea and vomiting in gynaecological patients undergoing laparoscopic surgery. Br J Anaesth. 2015 Dec;115(6):883-9. doi: 10.1093/bja/aev352. Epub 2015 Oct 27. PMID 26507494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Jan 2014 to Dec 2014 in North Institute of Huashan Hospital,Fudan University,Shanghai,China
Pre-assignment Details: 243 patients were assessed for eligibility, 86 were excluded for reasons below: Refused to participate. (n=12) Did not meet inclusion criteria. (n=71) Insufficient time to prepare for the study. (n=3)
Period: Overall Study
Arm/Group | Acustimulation | Tropisetron | Control
Started | 53 | 53 | 51
Completed | 50 | 53 | 50
Not Completed | 3 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — converted to open procedures | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acustimulation | Tropisetron | Control | Total
Number analyzed (Participants) | 50 | 53 | 50 | 153
Age, Continuous [Median (Full Range); unit: years] | 37 [24 to 60] | 35 [23 to 60] | 35 [22 to 60] | 35 [22 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 53 | 50 | 153
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 50 | 53 | 50 | 153
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 50 | 53 | 50 | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Postoperative Nausea and Vomiting in 24h Postoperatively
Description: the total number including nausea, retching and vomiting within 24h after operation
Time Frame: within 24h after operation
Measure: Number; unit: participants
Arm/Group | Acustimulation | Tropisetron | Control
Number analyzed (Participants) | 50 | 53 | 50
participants | 14 | 14 | 25
Statistical Analysis 1: Comparison: Acustimulation vs Tropisetron vs Control; Test type: Superiority or Other; p = 0.021, Chi-squared

2. Secondary Outcome: Number of Participants Experiencing Postoperative Nausea in 24h Postoperatively
Time Frame: within 24h after the operation
Measure: Number; unit: participants
Arm/Group | Acustimulation | Tropisetron | Control
Number analyzed (Participants) | 50 | 53 | 50
participants | 14 | 14 | 25
Statistical Analysis 1: Comparison: Acustimulation vs Tropisetron vs Control; Test type: Superiority or Other; p = 0.021, Chi-squared

3. Secondary Outcome: Number of Participants Experiencing Postoperative Vomiting in 24h Postoperatively
Description: including retching and vomiting
Time Frame: within 24h after operation
Measure: Number; unit: participants
Arm/Group | Acustimulation | Tropisetron | Control
Number analyzed (Participants) | 50 | 53 | 50
participants | 9 | 8 | 12
Statistical Analysis 1: Comparison: Acustimulation vs Tropisetron vs Control; Test type: Superiority or Other; p = 0.503, Chi-squared

4. Other Pre Specified Outcome: Need of Postoperative Metoclopramide
Description: the number of patients who needed metoclopramide as a rescue medicine postoperatively
Time Frame: within 48h after operation
Measure: Number; unit: participants
Arm/Group | Acustimulation | Tropisetron | Control
Number analyzed (Participants) | 50 | 53 | 50
participants | 5 | 4 | 7
Statistical Analysis 1: Comparison: Acustimulation vs Tropisetron vs Control; Test type: Superiority or Other; p = 0.571, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the start of anesthesia to 48h after the operation.
Arm/Group | Acustimulation | Tropisetron | Control
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/51
Other Adverse Events (participants affected / at risk) | 6/53 | 0/53 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acustimulation (N=53) | Tropisetron (N=53) | Control (N=51)
Local redness (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Local itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Local skin swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes